CLINICAL TRIAL: NCT02121795
Title: A Phase 3, Randomized, Double-Blind, Switch Study to Evaluate F/TAF in HIV-1 Positive Subjects Who Are Virologically Suppressed on Regimens Containing FTC/TDF
Brief Title: Switch Study to Evaluate F/TAF in HIV-1 Positive Participants Who Are Virologically Suppressed on Regimens Containing FTC/TDF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-311-1089; 2013-005138-39 (EudraCT Number)
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: HIV-1 Infection
Keywords: HIV; HIV-1 Positive; Virologically-suppressed
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- F/TAF + 3rd Agent (Experimental): Participants will receive F/TAF (200/25 mg or 200/10 mg) plus FTC/TDF placebo while remaining on an allowed third antiretroviral agent of the participant's pre-existing treatment regimen, for 96 weeks. Dosing of F/TAF will be dependent on the third agent of the participants' pre-existing treatment regimen.
  Interventions: Drug: F/TAF; Drug: Allowed third antiretroviral agent; Drug: FTC/TDF Placebo
- FTC/TDF + 3rd Agent (Active Comparator): Participants will receive FTC/TDF plus F/TAF placebo while remaining on an allowed third antiretroviral agent of the participant's pre-existing treatment regimen, for 96 weeks.
  Interventions: Drug: FTC/TDF; Drug: Allowed third antiretroviral agent; Drug: F/TAF Placebo

INTERVENTIONS:
Drug: FTC/TDF — 200/300 mg FDC tablets administered orally once daily
  Other Names: Truvada®
  Arms: FTC/TDF + 3rd Agent
Drug: F/TAF — Tablets administered orally once daily
  Other Names: Descovy®
  Arms: F/TAF + 3rd Agent
Drug: Allowed third antiretroviral agent — An allowed third antiretroviral agent of the participant's pre-existing regimen may include one of the following: ritonavir-boosted atazanavir (ATV/r), ritonavir-boosted lopinavir (LPV/r), ritonavir-boosted darunavir (DRV/r), efavirenz (EFV; Sustiva®), rilpivirine (RPV; Edurant®), nevirapine (NVP;Viramune®), raltegravir (RAL; Isentress®), dolutegravir (DTG;Tivicay®), and maraviroc (MVC; Selzentry®).
Drug: FTC/TDF Placebo — Tablets administered orally once daily
  Arms: F/TAF + 3rd Agent
Drug: F/TAF Placebo — Tablets administered orally once daily
  Arms: FTC/TDF + 3rd Agent

SUMMARY:
This study will evaluate the efficacy of switching from emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) fixed dose combination (FDC) to emtricitabine/tenofovir alafenamide (F/TAF) FDC in HIV-1 positive participants who are virologically suppressed on regimens containing FTC/TDF.

This study will consist of a 96 week double-blind treatment period. After Week 96, all participants will continue on blinded study drug treatment and attend visits every 12 weeks until treatment assignments are unblinded. All participants will return for an unblinding visit and will be given the option to receive open-label F/TAF and attend visits every 12 weeks until F/TAF is commercially available, or the sponsor terminates the F/TAF clinical development program.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Currently receiving antiretroviral regimen containing FTC/TDF in combination with one third agent for ≥ 6 consecutive months prior to screening.
* Plasma HIV-1 RNA levels < 50 copies/mL for at least 6 months preceding the screening visit (measured at least twice using the same assay) and not experienced two consecutive HIV-1 RNA above detectable levels after achieving a confirmed (two consecutive) HIV-1 RNA below detectable levels on the current regimen in the past year.
* Plasma HIV-1 RNA should be < 50 copies/mL at the screening visit.
* Normal electrocardiogram (ECG)
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min according to the Cockcroft-Gault formula for creatinine clearance
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × the upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin (individuals with documented Gilbert's syndrome or with Atazanavir-associated hyperbilirubinemia may have total bilirubin up to 5 x ULN)
* Adequate hematologic function
* Serum amylase ≤ 5 × ULN
* Females of childbearing potential must agree to utilize highly effective contraception methods or be non-heterosexually active, or practice abstinence from screening throughout the duration of the study treatment and for 30 days following the last dose of the study drug.
* Females who have stopped menstruating for ≥ 12 months but do not have documentation of ovarian hormonal failure must have a serum follicle stimulating hormone (FSH) level at screening within the post-menopausal range based on the Central Laboratory reference range.
* Females who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing.
* Males must agree to utilize a highly effective method of contraception during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence from first dose throughout the study period and for 30 days following the last study drug dose.

Key Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Hepatitis C virus (HCV) antibody positive and HCV RNA detectable
* Individuals experiencing decompensated cirrhosis (e.g., ascites, encephalopathy, etc.)
* Individuals receiving ongoing treatment with bisphosphonate to treat bone disease (eg, osteoporosis)
* Females who are breastfeeding
* Positive serum pregnancy test
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the investigator to potentially interfere with study compliance
* A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1 Visit
* Individuals receiving ongoing therapy with any of the medications not to be used with FTC, TAF, TDF or other antiretroviral third agents.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2014-05-06 (Actual); Primary Completion 2015-08-12 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (78):
- United States (57):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Kaiser Permanente, Hayward, California
  - Tarrant County ID Associates, Los Angeles, California
  - Southern California Men's Medical Group, Los Angeles, California
  - Highland Hospital - Alameda Health System (formerly Alameda County medical Center), Oakland, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Kaiser Permanente Medical Group San Francisco, San Francisco, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Kaiser Permanente Colorado, Denver, Colorado
  - National Jewish Health, Denver, Colorado
  - Apex Research LLC, Denver, Colorado
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Capital Medical Associates, Washington D.C., District of Columbia
  - Medical Faculty Associates, Washington D.C., District of Columbia
  - TheraFirst Medical Center, Fort Lauderdale, Florida
  - Gary J. Richmond,M.D.,P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Tarrant County Infectious Disease Associates, Miami, Florida
  - AIDS Healthcare Foundation, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - AIDS Healthcare Foundation, Tampa, Florida
  - AIDS Research & Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Atlanta ID Group, Atlanta, Georgia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Community Research Initiative of New England, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - The Kc Care Clinic Site 5580, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Prime Healthcare Services - St Michael's LLC d/b/a Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - New York Hospital Queens, Flushing, New York
  - North Shore University Hospital, Manhasset, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Infectious Disease Consultants, PA, Charlotte, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Central Texas Clinical Research, Austin, Texas
  - AIDS Arms, Inc, Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Inc, Dallas, Texas
  - North Texas Infectious Diseases Consulants, Dallas, Texas
  - AIDS Arms, Inc./Trinity Health & Wellness Center, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Peter Shalit, MD, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- CHU Saint-Pierre of Brussels, Brussels, Belgium
- Canada (4):
  - Vancouver Infectious Disease Research and Care Centre, Vancouver, British Columbia
  - Ottawa Hospital-General Campus, Ottawa, Ontario
  - Maple Leaf Medical Clinic/Maple Leaf Research, Toronto, Ontario
  - University Health Network/Toronto General Hospital, Toronto, Ontario
- France (5):
  - University Hospital of Montpellier (CHU-Gui de Chauliac), Montpellier
  - CHU de Nantes Hopital de l'Hotel Dieu, Nantes
  - Hopital Bichat Claude Bernard, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier de Tourcoing, Tourcoing
- Italy (2):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - IRCCS Ospedale San Raffaele, Centro San Luigi, Milan
- Puerto Rico (3):
  - Hope Clinical Research, San Juan
  - Clinical Research Puerto Rico Inc, San Juan
  - University of Puerto Rico School of Medicine, San Juan
- United Kingdom (6):
  - Brighton and Sussex University Hospitals, Brighton
  - Barts Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - King's College Hospital, London
  - Chelsea and Westminster Hospital, London
  - Manchester Centre for Sexual Health, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Derived] Gallant JE, Daar ES, Raffi F, Brinson C, Ruane P, DeJesus E, Johnson M, Clumeck N, Osiyemi O, Ward D, Morales-Ramirez J, Yan M, Abram ME, Plummer A, Cheng AK, Rhee MS. Efficacy and safety of tenofovir alafenamide versus tenofovir disoproxil fumarate given as fixed-dose combinations containing emtricitabine as backbones for treatment of HIV-1 infection in virologically suppressed adults: a randomised, double-blind, active-controlled phase 3 trial. Lancet HIV. 2016 Apr;3(4):e158-65. doi: 10.1016/S2352-3018(16)00024-2. Epub 2016 Mar 14. PMID 27036991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Europe. The first participant was screened on 06 May 2014. The last study visit occurred on 1 March 2019.
Pre-assignment Details: 780 participants were screened.
Groups:
- F/TAF + 3rd Agent: Double-Blind Phase: emtricitabine/tenofovir alafenamide (F/TAF) (200/25 mg or 200/10 mg) tablet + emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) placebo tablet + third agent administered orally once daily for at least 96 weeks.
  Open-Label Phase: After Week 96, participants continued to take their blinded study drug and attended visits every 12 weeks until treatment assignments were unblinded, at which point all participants returned for an unblinding visit and were given the option to receive open-label F/TAF and attend visits every 12 weeks until F/TAF was commercially available or until Gilead Sciences terminated the F/TAF clinical development program.
- FTC/TDF + 3rd Agent: Double-Blind Phase: FTC/TDF 200/300 mg tablet + F/TAF placebo tablet + third agent administered orally once daily for at least 96 weeks.
  Open-Label Phase: After Week 96, participants continued to take their blinded study drug and attended visits every 12 weeks until treatment assignments were unblinded, at which point all participants returned for an unblinding visit and were given the option to receive open-label F/TAF and attend visits every 12 weeks until F/TAF was commercially available or until Gilead Sciences terminated the F/TAF clinical development program.
Period: Double-Blind Phase
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Started | 334 | 334
Safety Analysis Set | 333 | 330
Completed | 296 | 300
Not Completed | 38 | 34
Not completed — Randomized but Never Treated | 1 | 4
Not completed — Withdrawal by Subject | 19 | 16
Not completed — Lost to Follow-up | 7 | 4
Not completed — Physician Decision | 2 | 5
Not completed — Adverse Event | 5 | 0
Not completed — Non-Compliance with Study Drug | 3 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Death | 1 | 1
Period: Open-Label Phase
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Started | 33 (Not all participants entered the Open-Label Phase.) | 31 (Not all participants entered the Open-Label Phase.)
Completed | 21 | 21
Not Completed | 12 | 10
Not completed — Physician Decision | 8 | 8
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study drug.
Groups:
- F/TAF + 3rd Agent: Double-Blind Phase: F/TAF (200/25 mg or 200/10 mg) tablet + emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) placebo tablet + third agent administered orally once daily for at least 96 weeks.
- FTC/TDF + 3rd Agent: Double-Blind Phase: FTC/TDF 200/300 mg tablet + F/TAF placebo tablet + third agent administered orally once daily for at least 96 weeks.
- Total: Total of all reporting groups
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent | Total
Number analyzed (Participants) | 333 | 330 | 663
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47 (9.9) | 48 (9.7) | 48 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 54 | 102
  Male | 285 | 276 | 561
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 78 | 126
  Not Hispanic or Latino | 285 | 252 | 537
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 6 | 0 | 6
  Black | 69 | 67 | 136
  Native Hawaiian or Pacific Islander | 2 | 1 | 3
  White | 244 | 253 | 497
  Not Permitted | 1 | 1 | 2
  Other | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 9 | 14
  Belgium | 3 | 3 | 6
  United States | 282 | 274 | 556
  Italy | 2 | 6 | 8
  United Kingdom | 23 | 17 | 40
  France | 18 | 21 | 39
Baseline Third Agent [Number; unit: participants]
  Atazanavir boosted with ritonavir (ATV/r) | 53 | 50 | 103
  Darunavir boosted with ritonavir (DRV/r) | 84 | 82 | 166
  Lopinavir boosted with ritonavir (LPV/r) | 18 | 18 | 36
  Dolutegravir (DTG) | 26 | 23 | 49
  Efavirenz (EFV) | 8 | 6 | 14
  Maraviroc (MVC) | 1 | 6 | 7
  Nevirapine (NVP) | 74 | 66 | 140
  Raltegravir (RAL) | 66 | 73 | 139
  Rilpivirine (RPV) | 3 | 6 | 9
HIV-1 RNA Categories [Number; unit: participants]
  < 50 copies/mL | 329 | 326 | 655
  >= 50 copies/mL | 4 | 4 | 8
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 691 (272.6) | 667 (272.3) | 679 (272.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the FDA Snapshot Analysis
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: The Full Analysis Set included all participants who were randomized into the study and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 333 | 330
percentage of participants | 94.3 | 93.0
Statistical Analysis 1: Comparison: F/TAF + 3rd Agent vs FTC/TDF + 3rd Agent; Test type: Non-Inferiority — Noninferiority was assessed using a conventional 95.002% confidence interval (CI) approach, with a noninferiority margin of 10%; p = 0.5, Cochran-Mantel-Haenszel; P-value was from Cochran-Mantel-Haenszel (CMH) test stratified by third agent; Percentage difference = 1.3, 95.002% CI 2-sided [-2.5 to 5.1] — Difference in percentages of virologic success between treatment groups and its 95.002% CI were calculated based on the Mantel-Haenszel (MH) proportions adjusted by the third agent stratum

2. Secondary Outcome: Percentage Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Description: Hip BMD was assessed by dual energy x-ray absorptiometry (DXA) scan.
Time Frame: Baseline; Week 48
Population: Participants in the Hip DXA Analysis Set (participants who were randomized and received at least one dose of study drug and had nonmissing baseline hip BMD data) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 304 | 305
percentage change | 1.236 (2.6602) | -0.071 (2.3316)

3. Secondary Outcome: Percentage Change From Baseline in Spine BMD at Week 48
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set (participants who were randomized and received at least one dose of study drug and had nonmissing baseline spine BMD data) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 304 | 309
percentage change | 1.662 (3.1279) | -0.109 (3.3476)

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 48 as Defined by the FDA Snapshot Analysis
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 333 | 330
percentage of participants | 91.6 | 90.9

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 313 | 311
cells/μL | 20 (161.8) | 21 (152.7)

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 96 as Defined by the FDA Snapshot Analysis
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 333 | 330
percentage of participants | 83.5 | 86.1

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Weeks 96 as Defined by the FDA Snapshot Analysis
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 333 | 330
percentage of participants | 88.6 | 89.1

8. Secondary Outcome: Percentage Change From Baseline in Hip BMD at Week 96
Description: Hip BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 291 | 292
percentage change | 1.856 (3.2195) | -0.289 (2.9912)

9. Secondary Outcome: Percentage Change From Baseline in Spine BMD at Week 96
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 290 | 296
percentage change | 2.159 (3.8374) | -0.109 (3.6738)

10. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | F/TAF + 3rd Agent | FTC/TDF + 3rd Agent
Number analyzed (Participants) | 299 | 296
cells/μL | 50 (198.7) | 46 (169.4)

ADVERSE EVENTS:
Time Frame: First dose of study drug to the last dose (maximum: 227.4 weeks) plus 30 days
Description: The Safety Analysis Set included all randomized participants who received at least one dose of study drug.
Groups:
- F/TAF + 3rd Agent (Double-Blind): Double-Blind Phase: F/TAF (200/25 mg or 200/10 mg tablet) + FTC/TDF placebo tablet + third agent administered orally once daily for at least 96 weeks.
- FTC/TDF + 3rd Agent (Double-Blind): Double-Blind Phase: FTC/TDF 200/300 mg tablet + F/TAF placebo tablet + third agent administered orally once daily for at least 96 weeks.
- Open-Label F/TAF From F/TAF: Open-Label Phase: F/TAF (200/25 mg or 200/10 mg) tablet orally once daily until F/TAF was commercially available or until Gilead Sciences terminated the F/TAF clinical development program in participants from the F/TAF + 3rd Agent group.
- Open-Label F/TAF From FTC/TDF: Open-Label Phase: F/TAF (200/25 mg or 200/10 mg) tablet orally once daily until F/TAF was commercially available or until Gilead Sciences terminated the F/TAF clinical development program in participants from the FTC/TDF + 3rd Agent group.
Arm/Group | F/TAF + 3rd Agent (Double-Blind) | FTC/TDF + 3rd Agent (Double-Blind) | Open-Label F/TAF From F/TAF | Open-Label F/TAF From FTC/TDF
All-Cause Mortality (participants affected / at risk) | 2/333 | 1/330 | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 29/333 | 31/330 | 2/33 | 3/31
Other Adverse Events (participants affected / at risk) | 242/333 | 226/330 | 12/33 | 13/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | F/TAF + 3rd Agent (Double-Blind) (N=333) | FTC/TDF + 3rd Agent (Double-Blind) (N=330) | Open-Label F/TAF From F/TAF (N=33) | Open-Label F/TAF From FTC/TDF (N=31)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 1 | 1 | 0
Drowning (General disorders) | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Acute hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Bone tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Mycobacterium abscessus infection (Infections and infestations) | 1 | 0 | 0 | 0
Oesophagitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 0
Prostatitis Escherichia coli (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness exertional (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | F/TAF + 3rd Agent (Double-Blind) (N=333) | FTC/TDF + 3rd Agent (Double-Blind) (N=330) | Open-Label F/TAF From F/TAF (N=33) | Open-Label F/TAF From FTC/TDF (N=31)
Diarrhoea (Gastrointestinal disorders) | 44 | 42 | 1 | 0
Nausea (Gastrointestinal disorders) | 23 | 19 | 0 | 0
Fatigue (General disorders) | 26 | 23 | 0 | 0
Influenza like illness (General disorders) | 6 | 10 | 0 | 2
Pyrexia (General disorders) | 6 | 17 | 0 | 0
Bronchitis (Infections and infestations) | 32 | 26 | 1 | 1
Fungal skin infection (Infections and infestations) | 1 | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 11 | 8 | 2 | 0
Influenza (Infections and infestations) | 23 | 15 | 0 | 2
Nasopharyngitis (Infections and infestations) | 43 | 27 | 4 | 2
Onychomycosis (Infections and infestations) | 6 | 3 | 0 | 3
Sinusitis (Infections and infestations) | 23 | 28 | 2 | 3
Syphilis (Infections and infestations) | 18 | 7 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 54 | 67 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 23 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 28 | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 22 | 0 | 0
Headache (Nervous system disorders) | 33 | 22 | 0 | 1
Anxiety (Psychiatric disorders) | 15 | 20 | 2 | 1
Insomnia (Psychiatric disorders) | 15 | 13 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 20 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 19 | 11 | 1 | 0
Hypertension (Vascular disorders) | 16 | 20 | 0 | 0

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years